CLINICAL TRIAL: NCT05041907
Title: Finding Treatments for COVID-19: A Phase 2 Multi-centre Adaptive Platform Trial to Assess Antiviral Pharmacodynamics in Early Symptomatic COVID-19 (PLATCOV)
Brief Title: Finding Treatments for COVID-19: A Trial of Antiviral Pharmacodynamics in Early Symptomatic COVID-19 (PLATCOV)
Acronym: PLATCOV
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIR21001
Record Dates: First submitted 2021-09-07; First posted 2021-09-13 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: COVID-19
Keywords: COVID-19; Phase 2; Antiviral Pharmacodynamics
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir; Ritonavir; nitazoxanide; molnupiravir; Hydroxychloroquine; Antibodies, Monoclonal; Fluoxetine; sotrovimab; ensitrelvir; favipiravir; Ivermectin; remdesivir; Metformin; nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (19):
- Positive control: Nirmatrelvir/ritonavir (e.g. PAXLOVID™) (Active Comparator)
  Interventions: Drug: Nirmatrelvir/ritonavir (e.g. PAXLOVID™)
- Nitazoxanide (Experimental)
  Interventions: Drug: Nitazoxanide
- Molnupiravir and Nirmatrelvir/ritonavir (e.g. PAXLOVID™) [This arm is now closed to recruitment] (Experimental)
  Interventions: Drug: Molnupiravir and nirmatrelvir/ritonavir (e.g. PAXLOVID™)
- Hydroxychloroquine (Experimental)
  Interventions: Drug: Hydroxychloroquine
- Negative control group (Other)
  Interventions: Other: No treatment
- AZD7442 (EVUSHELD™) [This arm is now closed to recruitment] (Experimental)
  Interventions: Drug: Monoclonal antibodies
- Fluoxetine [This arm is now closed to recruitment] (Experimental)
  Interventions: Drug: Fluoxetine
- Molnupiravir [This arm is now closed to recruitment] (Experimental)
  Interventions: Drug: Molnupiravir
- Sotrovimab [Pending addition] (Experimental)
  Interventions: Drug: Sotrovimab
- Ensitrelvir [This arm is now closed to recruitment] (Experimental)
  Interventions: Drug: Ensitrelvir
- Positive control (REGN-COV2) [This arm is now closed to recruitment] (Active Comparator)
  Interventions: Drug: Monoclonal antibodies
- Favipiravir [This arm is now closed to recruitment] (Experimental)
  Interventions: Drug: Favipiravir
- Ivermectin [This arm is now closed to recruitment] (Experimental)
  Interventions: Drug: Ivermectin
- Remdesivir [This arm is now closed to recruitment] (Experimental)
  Interventions: Drug: Remdesivir
- Atilotrelvir/ritonavir [Pending addition] (Experimental)
  Interventions: Drug: Atilotrelvir/ritonavir
- Metformin (modified release) [Pending addition] (Experimental)
  Interventions: Drug: Metformin
- Nirmatrelvir/ritonavir - 300/50 - dose finding [Pending addition] (Experimental)
  Interventions: Drug: Nirmatrelvir/ritonavir
- Nirmatrelvir/ritonavir - 150/50 - dose finding [Pending addition] (Experimental)
  Interventions: Drug: Nirmatrelvir/ritonavir
- Nirmatrelvir - dose finding [Pending addition] (Experimental)
  Interventions: Drug: Nirmatrelvir

INTERVENTIONS:
Drug: Nirmatrelvir/ritonavir (e.g. PAXLOVID™) — Nirmatrelvir 300mg BD for 5/7 Ritonavir 100mg BD for 5/7
  Arms: Positive control: Nirmatrelvir/ritonavir (e.g. PAXLOVID™)
Drug: Nitazoxanide — Nitazoxanide 1.5g BD 7/7
  Arms: Nitazoxanide
Drug: Molnupiravir and nirmatrelvir/ritonavir (e.g. PAXLOVID™) — Molnupiravir 800mg BD for 5/7, Nirmatrelvir 300mg BD for 5/7, Ritonavir 100mg BD for 5/7
  Arms: Molnupiravir and Nirmatrelvir/ritonavir (e.g. PAXLOVID™) [This arm is now closed to recruitment]
Drug: Hydroxychloroquine — Hydroxychloroquine 400mg D0 BD and 400MG OD for a further 6/7
  Arms: Hydroxychloroquine
Other: No treatment — No treatment (except antipyretics- paracetamol)
  Arms: Negative control group
Drug: Monoclonal antibodies — Monoclonal antibodies: 300mg tixagevimab/ 300 mg cilgavimab given once on D0
  Arms: AZD7442 (EVUSHELD™) [This arm is now closed to recruitment]
Drug: Fluoxetine — Fluoxetine 40mg OD for 7/7
  Arms: Fluoxetine [This arm is now closed to recruitment]
Drug: Molnupiravir — Molnupiravir 800mg BD for 5/7
  Arms: Molnupiravir [This arm is now closed to recruitment]
Drug: Sotrovimab — Sotrovimab 500mg given once on D0
  Arms: Sotrovimab [Pending addition]
Drug: Ensitrelvir — Ensitrelvir 375mg OD D0 and 125mg OD for a further 4/7
  Arms: Ensitrelvir [This arm is now closed to recruitment]
Drug: Monoclonal antibodies — Monoclonal antibodies: 600mg casirivimab/ 600mg imdevimab given once on D0
  Arms: Positive control (REGN-COV2) [This arm is now closed to recruitment]
Drug: Favipiravir — Favipiravir 1800mg BD D0 and 800mg BD for a further 6/7
  Arms: Favipiravir [This arm is now closed to recruitment]
Drug: Ivermectin — Ivermectin 600micrograms/kg/day for 7/7.
  Arms: Ivermectin [This arm is now closed to recruitment]
Drug: Remdesivir — Remdesivir 200mg D0 and 100mg for a further 4/7.
  Arms: Remdesivir [This arm is now closed to recruitment]
Drug: Atilotrelvir/ritonavir — Atilotrelvir 150mg BD for 5/7 Ritonavir 100mg BD for 5/7
  Arms: Atilotrelvir/ritonavir [Pending addition]
Drug: Metformin — Metformin 500mg TDS 5/7
  Arms: Metformin (modified release) [Pending addition]
Drug: Nirmatrelvir/ritonavir — Nirmatrelvir 300mg BD for 5/7 Ritonavir 50mg BD for 5/7
  Arms: Nirmatrelvir/ritonavir - 300/50 - dose finding [Pending addition]
Drug: Nirmatrelvir/ritonavir — Nirmatrelvir 150mg BD for 5/7 Ritonavir 50mg BD for 5/7
  Arms: Nirmatrelvir/ritonavir - 150/50 - dose finding [Pending addition]
Drug: Nirmatrelvir — Nirmatrelvir 300mg BD for 5/7
  Arms: Nirmatrelvir - dose finding [Pending addition]

SUMMARY:
The trial will develop and validate a platform for quantitative assessment of antiviral effects in low-risk patients with high viral burdens and uncomplicated COVID-19 to determine in-vivo antiviral activity. In this randomized open label, controlled, group sequential adaptive platform trial, we will assess the performance of three distinct types of intervention relative to control (no treatment):

A: Small molecule drugs; B: Monoclonal antibodies; C: Dose finding for the constituent parts of nirmatrelvir/ritonavir

PLATCOV study is supported by the Wellcome Trust Grant ref: 223195/Z/21/Z through the COVID-19 Therapeutics Accelerator.

DETAILED DESCRIPTION:
The platform trial will assess drugs with potential SARS-CoV-2 antiviral activity of three general types:

A. Small molecule drugs: currently nitazoxanide, nirmatrelvir/ritonavir, hydroxychloroquine, atilotrelvir/ritonavir and metformin.

B. Monoclonal antibodies: Sotrovimab and any other monoclonal antibodies that become available. Monoclonal antibodies are vulnerable to viral escape mutations. Tracking their performance over time is important to characterise the impact and inform the therapeutics of mutant SARS-CoV-2 strains. This will also be important for other antivirals. Monoclonal antibodies are expensive and cannot be produced at large scale currently, but this may change in the near future. These drugs will be included if there is local availability and regulatory approval.

C. : Dose finding for the constituent parts of nirmatrelvir/ritonavir. Nirmatrelvir/ritonavir has shown clinical efficacy in phase III studies, however, there are disadvantages to using it (drug-drug interactions, side effects, cost). In the urgent context of the pandemic, a higher dose of ritonavir was chosen to guarantee maximum boosting effect. We do not know if the maximal boosting effect could have been achieved with less, or even without ritonavir. It will be investigated whether reducing the doses of the constituent parts can still retain the effectiveness.

Randomization to the no antiviral treatment control arm (no intervention) will be fixed at a minimum of 20% throughout the study. The randomization ratios will be uniform for all available interventions.

Recruitment into the ivermectin arm was stopped on April 18th 2022 due to meeting the pre- defined stopping criteria.

Recruitment into the remdesivir arm was stopped on June 10th 2022 due to meeting the pre- defined stopping criteria.

Recruitment into the REGN-COV2 arm was stopped on October 20th 2022 due to meeting the pre-defined stopping criteria.

Recruitment into the favipiravir arm was stopped on October 31st 2022 due to meeting the pre-defined stopping criteria.

Recruitment into the molnupiravir arm was stopped on February 22nd 2023 due to meeting the pre-defined stopping criteria.

Recruitment into the fluoxetine arm was stopped on May 8th 2023 due to meeting the pre-defined stopping criteria.

Recruitment into the evusheld arm was stopped on July 4th 2023 due to meeting the pre-defined stopping criteria.

Recruitment into the ensitrelvir arm was stopped on April 21st 2024 due to meeting the pre-defined stopping criteria.

Recruitment into the combination molnupiravir and nirmatrelvir/ritonavir (e.g. PAXLOVID™) arm was stopped on May 31st 2024 due to meeting the pre-defined stopping criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patient understands the procedures and requirements and is willing and able to give informed consent for full participation in the study.
* Previously healthy adults, male or female, aged 18 to 60 years at time of consent with early symptomatic COVID-19
* SARS-CoV-2 positive by lateral flow antigen test OR a positive PCR test for SARS-CoV-2 within the last 24hrs with a Ct value of less than 25 (all viral targets)
* Symptoms of COVID-19 (including fever, or history of fever) for less than 4 days (96 hours).
* Oxygen saturation ≥96% measured by pulse-oximetry at time of screening.
* Able to walk unaided and unimpeded in ADLs
* Agrees and is able to adhere to all study procedures, including availability and contact information for follow-up visits

Exclusion Criteria:

The patient may not enter the study if ANY of the following apply:

* Taking any concomitant medications or drugs (see appendix 4)†
* Presence of any chronic illness/ condition requiring long term treatment, or other significant comorbidity (e.g. diabetes, obesity but see appendix 4 for the full list)
* Laboratory abnormalities discovered at screening (see appendix 4)
* For females: pregnancy, actively trying to become pregnant, or lactation
* Contraindication to taking, or known hypersensitivity reaction to any of the proposed therapeutics (see appendix 4)
* Currently participating in another COVID-19 therapeutic or vaccine trial
* Evidence of pneumonia (although imaging is NOT required)

  * healthy women on the oral contraceptive pill are eligible to join the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3800 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Rate of viral clearance for interventions relative to the no study arm (This is a superiority comparison) | Days 0-5
  Rate of viral clearance- estimated from the log10 viral density derived from qPCR of standardised duplicate oropharyngeal swabs/ saliva taken daily from baseline (day 0) to day 5 for each intervention compared with the no antiviral treatment control i.e., those not receiving study drug
Rate of viral clearance for interventions relative to the positive control arm (This is a non-inferiority or superiority comparison). | Days 0-5
  Rate of viral clearance- estimated from the log10 viral density derived from qPCR of standardised duplicate oropharyngeal swabs/ saliva taken daily from baseline (day 0) to day 5 for interventions compared with the current best antiviral treatment option (accelerated viral clearance relative to the positive control arm)

SECONDARY OUTCOMES:
Viral kinetic levels in early COVID-19 disease | Days 0-5
  Rate of viral clearance estimated from the log10 viral density derived from qPCR of standardised duplicate oropharyngeal swabs/ saliva taken daily from baseline (day 0) to day 5 for each therapeutic arm compared with the no antiviral treatment control i.e., those not receiving study drug
Optimal dosing regimens through pharmacometric assessment for antiviral drugs with evidence of efficacy in the literature or from the trial data (e.g., Nirmatrelvir/ritonavir, Ensitrelvir etc). | Days 0-5
  Rate of viral clearance- estimated from the log10 viral density derived from qPCR of standardised duplicate oropharyngeal swabs/ saliva taken daily from baseline (day 0) to day 5 for each therapeutic arm compared with the no antiviral treatment control i.e., those not receiving study drug
Viral rebound of studied treatment arms in comparison to contemporaneous controls (e.g. no study drug arm, positive control) | Days 6-14
  After stopping treatment for at least 24 hours (or 5 days if no drug is given or a single dose monoclonal antibody is given), rebound is defined as an oropharyngeal eluate viral density estimate >1000 genomes per ml for at least 1 timepoint (average 2 swabs), after >2 consecutive days of average daily viral density estimate less than 100 genomes per ml
Rates of fever clearance and symptom resolution with respect to no treatment | Days 0-14
  The following endpoints will be used:
  * Time to resolution of fever
  * Area Under the Curve of recorded temperature
  * Time to resolution of symptoms

OTHER OUTCOMES:
Rates of hospitalisation by treatment arm (hospitalisation for clinical reasons) | Days 0-28
  Number of hospitalisations up to Day 28 in a treatment arm with an increased rate of viral clearance compared with the negative control i.e. patients not receiving study drug
Relationship between viral clearance, randomisation arm and other measures (covariates) and development of post- acute COVID-19 (i.e. long COVID) | Days 0-120
  Score on post-acute COVID-19 (i.e. long COVID) questionnaire at day 120 - modified COVID-19 Yorkshire Rehabilitation Scale (C19 YRSm)

CONTACTS AND LOCATIONS:
Locations (7):
- Universidade Federal de Minas Gerais, Minas Gerais, Brazil
- Laos-Oxford-Mahosot Wellcome Trust Research Unit, Vientiane, Laos
- Sukraraj Tropical & Infectious Disease Hospital, Kathmandu, Nepal
- The Aga Khan University Hospital, Karachi, Pakistan
- Thailand (3):
  - Vajira hospital, Bangkok
  - Faculty of Tropical Medicine, Mahidol University, Bangkok
  - Bangplee Hospital, Mueang Samut Prakan

IPD SHARING:
Plan to Share IPD: Yes
With patient's consent, clinical data and results from blood analyses stored in the database may be shared according to the terms defined in the MORU data sharing policy with other researchers to use in the future.
  Data generated from this study will adhere to the 2016 "Statement on data sharing in public health emergencies"(https://wellcome.ac.uk/press-release/statement-data-sharing-public-health-emergencies).
Supporting Information: CSR, Analytic Code
Time Frame: after the main paper has been published
Access Criteria: MORU Data Sharing Policy https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing.
  The criteria for authorship will be consistent with the international guidelines (http://www.icmje.org/#author).
URL: http://wellcome.ac.uk/press-release/statement-data-sharing-public-health-emergencies

REFERENCES:
- [Derived] Kaewkhao N, Tarning J, Blessborn D. LC-MS/MS Method Validation for Quantification of Nirmatrelvir in Human Plasma. Int J Anal Chem. 2025 Nov 17;2025:6625833. doi: 10.1155/ianc/6625833. eCollection 2025. PMID 41321979
- [Derived] Schilling WHK, Jittamala P, Wongnak P, Watson JA, Boyd S, Luvira V, Siripoon T, Ngamprasertchai T, Batty EM, Beer E, Singh S, Asawasriworanan T, Seers T, Phommasone K, Evans TJ, Kruabkontho V, Ngernseng T, Tubprasert J, Abdad MY, Madmanee W, Kouhathong J, Suwannasin K, Pagornrat W, Piteekan T, Hanboonkunupakarn B, Poovorawan K, Potaporn M, Srisubat A, Loharjun B, Chotivanich K, Imwong M, Pukrittayakamee S, Dondorp AM, Day NPJ, Piyaphanee W, Phumratanaprapin W, White NJ; PLATCOV Collaborative Group. Antiviral efficacy of oral ensitrelvir versus oral ritonavir-boosted nirmatrelvir in COVID-19 (PLATCOV): an open-label, phase 2, randomised, controlled, adaptive trial. Lancet Infect Dis. 2025 Oct 10:S1473-3099(25)00482-7. doi: 10.1016/S1473-3099(25)00482-7. Online ahead of print. PMID 41082886
- [Derived] Jittamala P, Boyd S, Schilling WHK, Watson JA, Ngamprasertchai T, Siripoon T, Luvira V, Batty EM, Wongnak P, Esper LM, Almeida PJ, Cruz C, Ascencao FR, Aguiar RS, Ghanchi NK, Callery JJ, Singh S, Kruabkontho V, Ngernseng T, Tubprasert J, Madmanee W, Suwannasin K, Promsongsil A, Hanboonkunupakarn B, Poovorawan K, Potaporn M, Srisubat A, Loharjun B, Taylor WRJ, Qamar F, Kazi AM, Beg MA, Chommanam D, Vidhamaly S, Chotivanich K, Imwong M, Pukrittayakamee S, Dondorp AM, Day NPJ, Teixeira MM, Piyaphanee W, Phumratanaprapin W, White NJ; PLATCOV Collaborative Group. Antiviral efficacy of fluoxetine in early symptomatic COVID-19: an open-label, randomised, controlled, adaptive platform trial (PLATCOV). EClinicalMedicine. 2025 Jan 18;80:103036. doi: 10.1016/j.eclinm.2024.103036. eCollection 2025 Feb. PMID 39896880
- [Derived] Wongnak P, Schilling WHK, Jittamala P, Boyd S, Luvira V, Siripoon T, Ngamprasertchai T, Batty EM, Singh S, Kouhathong J, Pagornrat W, Khanthagan P, Hanboonkunupakarn B, Poovorawan K, Mayxay M, Chotivanich K, Imwong M, Pukrittayakamee S, Ashley EA, Dondorp AM, Day NPJ, Teixeira MM, Piyaphanee W, Phumratanaprapin W, White NJ, Watson JA; PLATCOV Collaborative Group. Temporal changes in SARS-CoV-2 clearance kinetics and the optimal design of antiviral pharmacodynamic studies: an individual patient data meta-analysis of a randomised, controlled, adaptive platform study (PLATCOV). Lancet Infect Dis. 2024 Sep;24(9):953-963. doi: 10.1016/S1473-3099(24)00183-X. Epub 2024 Apr 24. PMID 38677300
- [Derived] Luvira V, Schilling WHK, Jittamala P, Watson JA, Boyd S, Siripoon T, Ngamprasertchai T, Almeida PJ, Ekkapongpisit M, Cruz C, Callery JJ, Singh S, Tuntipaiboontana R, Kruabkontho V, Ngernseng T, Tubprasert J, Abdad MY, Keayarsa S, Madmanee W, Aguiar RS, Santos FM, Hanboonkunupakarn P, Hanboonkunupakarn B, Poovorawan K, Imwong M, Taylor WRJ, Chotivanich V, Chotivanich K, Pukrittayakamee S, Dondorp AM, Day NPJ, Teixeira MM, Piyaphanee W, Phumratanaprapin W, White NJ; PLATCOV Collaborative Group. Clinical antiviral efficacy of favipiravir in early COVID-19 (PLATCOV): an open-label, randomised, controlled, adaptive platform trial. BMC Infect Dis. 2024 Jan 15;24(1):89. doi: 10.1186/s12879-023-08835-3. PMID 38225598
- [Derived] Schilling WHK, Jittamala P, Watson JA, Boyd S, Luvira V, Siripoon T, Ngamprasertchai T, Batty EM, Cruz C, Callery JJ, Singh S, Saroj M, Kruabkontho V, Ngernseng T, Tanglakmankhong N, Tubprasert J, Abdad MY, Madmanee W, Kouhathong J, Suwannasin K, Pagornrat W, Piaraksa N, Hanboonkunupakarn P, Hanboonkunupakarn B, Poovorawan K, Potaporn M, Srisubat A, Loharjun B, Taylor WRJ, Chotivanich V, Chotivanich K, Imwong M, Pukrittayakamee S, Dondorp AM, Day NPJ, Teixeira MM, Piyaphanee W, Phumratanaprapin W, White NJ; PLATCOV Collaborative Group. Antiviral efficacy of molnupiravir versus ritonavir-boosted nirmatrelvir in patients with early symptomatic COVID-19 (PLATCOV): an open-label, phase 2, randomised, controlled, adaptive trial. Lancet Infect Dis. 2024 Jan;24(1):36-45. doi: 10.1016/S1473-3099(23)00493-0. Epub 2023 Sep 28. PMID 37778363
- [Derived] Jittamala P, Schilling WHK, Watson JA, Luvira V, Siripoon T, Ngamprasertchai T, Almeida PJ, Ekkapongpisit M, Cruz C, Callery JJ, Boyd S, Anunsittichai O, Hongsuwan M, Singhaboot Y, Pagornrat W, Tuntipaiboontana R, Kruabkontho V, Ngernseng T, Tubprasert J, Abdad MY, Keayarsa S, Madmanee W, Aguiar RS, Santos FM, Batty EM, Hanboonkunupakarn P, Hanboonkunupakarn B, Sookprome S, Poovorawan K, Imwong M, Taylor WRJ, Chotivanich V, Sangketchon C, Ruksakul W, Chotivanich K, Pukrittayakamee S, Dondorp AM, Day NPJ, Teixeira MM, Piyaphanee W, Phumratanaprapin W, White NJ; PLATCOV Collaborative Group. Clinical Antiviral Efficacy of Remdesivir in Coronavirus Disease 2019: An Open-Label, Randomized Controlled Adaptive Platform Trial (PLATCOV). J Infect Dis. 2023 Nov 11;228(10):1318-1325. doi: 10.1093/infdis/jiad275. PMID 37470445
- [Derived] Schilling WHK, Jittamala P, Watson JA, Ekkapongpisit M, Siripoon T, Ngamprasertchai T, Luvira V, Pongwilai S, Cruz C, Callery JJ, Boyd S, Kruabkontho V, Ngernseng T, Tubprasert J, Abdad MY, Piaraksa N, Suwannasin K, Hanboonkunupakarn P, Hanboonkunupakarn B, Sookprome S, Poovorawan K, Thaipadungpanit J, Blacksell S, Imwong M, Tarning J, Taylor WRJ, Chotivanich V, Sangketchon C, Ruksakul W, Chotivanich K, Teixeira MM, Pukrittayakamee S, Dondorp AM, Day NPJ, Piyaphanee W, Phumratanaprapin W, White NJ; PLATCOV Collaborative Group. Pharmacometrics of high-dose ivermectin in early COVID-19 from an open label, randomized, controlled adaptive platform trial (PLATCOV). Elife. 2023 Feb 21;12:e83201. doi: 10.7554/eLife.83201. PMID 36803992

DOCUMENTS (1):
  • Study Protocol (2024-08-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT05041907/Prot_001.pdf